CLINICAL TRIAL: NCT00610649
Title: Single Center, Randomized, Placebo-Controlled Trial to Establish Maximum Tolerated Dose, Optimal Titration Schedule, Safety, Tolerability, and Pharmacokinetics of Org 26576 in Patients Diagnosed With Major Depressive Disorder (Protocol No. P174001)
Brief Title: Trial to Determine the Maximum Tolerated Dose (MTD) Based on Safety and Tolerability, of Org 26576 in Participants With Major Depressive Disorder (174001/P05704/MK-8777-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05704; 174001 (Other: Organon Protocol Number)
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Depression
Keywords: randomized; placebo controlled; maximum tolerated dose
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part 1: Block A MK-8777 (Experimental): Participants receive MK-8777 initiated at 100 mg BID and titrated to a maximum of 600 mg BID. Participants receive MK-8777 for a total of 16 days.
  Interventions: Drug: MK-8777
- Part 1: Block A Placebo (Placebo Comparator): Participants receive placebo BID for a total of 16 days.
  Interventions: Drug: Placebo
- Part 1: Block B MK-8777 (Experimental): Participants receive MK-8777 initiated at 200 mg BID and titrated to a maximum of 600 mg BID. Participants receive MK-8777 for a total of 13 days.
  Interventions: Drug: MK-8777
- Part 1: Block B Placebo (Placebo Comparator): Participants receive placebo BID for a total of 13 days.
  Interventions: Drug: Placebo
- Part 1: Block C MK-8777 (Experimental): Participants receive MK-8777 initiated at 300 mg BID and titrated to a maximum of 600 mg BID. Participants receive MK-8777 for a total of 10 days.
  Interventions: Drug: MK-8777
- Part 1: Block C Placebo (Placebo Comparator): Participants receive placebo BID for a total of 10 days.
  Interventions: Drug: Placebo
- Part 1: Block D MK-8777 (Experimental): Participants receive MK-8777 initiated at 100 mg BID and titrated to a maximum dose determined by the results of Block A. Participants receive MK-8777 for a total of 13 days.
  Interventions: Drug: MK-8777
- Part 1: Block D Placebo (Placebo Comparator): Participants receive placebo BID for a total of 13 days.
  Interventions: Drug: Placebo
- Part 2: MK-8777 200 mg (Experimental): Participants receive MK-8777 100 mg BID for 27 days followed by one day of 100 mg QD. Participants receive MK-8777 for a total of 28 days.
  Interventions: Drug: MK-8777
- Part 2: MK-8777 800 mg (Experimental): Participants receive MK-8777 200 mg BID for 3 days followed by 400 mg BID for 24 days followed by one day of 400 mg QD. Participants receive MK-8777 for a total of 28 days.
  Interventions: Drug: MK-8777
- Part 2: Placebo (Placebo Comparator): Participants receive placebo BID for 27 days followed by one day of placebo QD. Participants receive placebo for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8777 — Orally administered capsules containing either 50 mg or 100 mg MK-8777.
  Arms: Part 1: Block A MK-8777; Part 1: Block B MK-8777; Part 1: Block C MK-8777; Part 1: Block D MK-8777; Part 2: MK-8777 200 mg; Part 2: MK-8777 800 mg
Drug: Placebo — Orally administered matching placebo capsules.
  Arms: Part 1: Block A Placebo; Part 1: Block B Placebo; Part 1: Block C Placebo; Part 1: Block D Placebo; Part 2: Placebo

SUMMARY:
Trial to determine the maximum tolerated dose (MTD) based on safety and tolerability of MK-8777 (Org 26576, SCH 900777) in participants with major depressive disorder.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, safety and tolerability study examining MK-8777 in participants with major depressive disorder. In Part I of the trial, four different cohorts of six participants each will receive multiple rising doses of MK-8777 (ranging from 100 mg twice a day [BID] to 300 mg BID) or placebo for up to 16 days. In Part 2, a new cohort of participants will be randomly assigned to receive 100 mg BID of MK-8777, 400 mg BID of MK-8777, or placebo. Following titration (3 days per step), participants will be maintained on the assigned BID dose until Day 27, followed by one day of once a day (QD) dosing, for a total of 28 days. There were 11 treatment arms in total for Part 1 and Part 2 (see Interventions).

ELIGIBILITY:
Inclusion Criteria:

* Female who is non-pregnant, nonlactating, using an acceptable method of birth control, or is not of child-bearing potential;
* be diagnosed with current major depressive disorder either mild or severe, as evidenced by a score of at least 9 but not more than 20 on the Quick Inventory of Depression Symptomatology - Clinician Rated (QIDS-C);
* be anti-depressant naïve;
* be able to refrain from all use of grapefruit containing products from the time of admission until the last assessment is performed at discharge;
* smokes less than or equal to 10 cigarettes or equivalent daily.

Exclusion Criteria:

* has any current and primary Axis I disorder other than major depressive disorder;
* has any history of bipolar I or II disorder, dysthymia, psychotic depression, psychotic disorders, posttraumatic stress disorder, borderline personality disorder, obsessive compulsive disorder, or eating disorder;
* the duration of the current depressive episode is longer than 2 years at screening;
* has any history of a significant suicide attempt, or poses a current risk of attempting suicide;
* is known to be human immunodeficiency virus (HIV) positive, or positive for hepatitis B surface antigen or hepatitis A antibodies or hepatitis C total antibodies;
* has any clinically significant concurrent endocrine, renal, respiratory, cardiovascular, hematological, immunological, cerebrovascular, neurological, malignancy, or any other concurrent medical condition, or has any history of diabetes mellitus;
* donation of blood within 60 days prior to the anticipated first dose of trial medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-09-20 (Actual); Primary Completion 2008-11-18 (Actual); Study Completion 2008-12-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Nations KR, Dogterom P, Bursi R, Schipper J, Greenwald S, Zraket D, Gertsik L, Johnstone J, Lee A, Pande Y, Ruigt G, Ereshefsky L. Examination of Org 26576, an AMPA receptor positive allosteric modulator, in patients diagnosed with major depressive disorder: an exploratory, randomized, double-blind, placebo-controlled trial. J Psychopharmacol. 2012 Dec;26(12):1525-39. doi: 10.1177/0269881112458728. Epub 2012 Sep 6. PMID 22954616

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Block A MK-8777: Participants receive MK-8777 initiated at 100 mg twice daily (BID) and titrated to a maximum of 600 mg BID. Participants receive MK-8777 for a total of 16 days.
- Part 2: MK-8777 200 mg: Participants receive MK-8777 100 mg BID for 27 days followed by one day of 100 mg once daily (QD). Participants receive MK-8777 for a total of 28 days.
Period: Overall Study
Arm/Group | Part 1: Block A MK-8777 | Part 1: Block A Placebo | Part 1: Block B MK-8777 | Part 1: Block B Placebo | Part 1: Block C MK-8777 | Part 1: Block C Placebo | Part 1: Block D MK-8777 | Part 1: Block D Placebo | Part 2: MK-8777 200 mg | Part 2: MK-8777 800 mg | Part 2: Placebo
Started | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2 | 10 | 10 | 10
Completed | 3 | 1 | 4 | 2 | 4 | 2 | 4 | 2 | 10 | 9 | 9
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Family Emergency | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Block A MK-8777 | Part 1: Block A Placebo | Part 1: Block B MK-8777 | Part 1: Block B Placebo | Part 1: Block C MK-8777 | Part 1: Block C Placebo | Part 1: Block D MK-8777 | Part 1: Block D Placebo | Part 2: MK-8777 200 mg | Part 2: MK-8777 800 mg | Part 2: Placebo | Total
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2 | 10 | 10 | 10 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (5.0) | 32.5 (13.4) | 42.0 (14.8) | 28.5 (9.2) | 35.5 (9.7) | 39.0 (14.1) | 40.5 (6.8) | 36.5 (23.3) | 38.3 (14.4) | 35.6 (12.8) | 31.1 (6.5) | 35.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 4 | 4 | 5 | 20
  Male | 4 | 2 | 0 | 1 | 2 | 2 | 4 | 2 | 6 | 6 | 5 | 34

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Moderate Intensity Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. A moderate intensity AE is defined as an AE that causes no significant interference with functioning.
Time Frame: Up to 7 days following the last dose of study drug (Up to 23 days)
Population: The All Subjects Treated (AST) population consisted of all Part 1 participants who received at least one dose of study drug (MK-8777 or Placebo).
Measure: Number; unit: participants
Arm/Group | Part 1: Block A MK-8777 | Part 1: Block A Placebo | Part 1: Block B MK-8777 | Part 1: Block B Placebo | Part 1: Block C MK-8777 | Part 1: Block C Placebo | Part 1: Block D MK-8777 | Part 1: Block D Placebo
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
participants | 2 | 0 | 1 | 2 | 4 | 0 | 3 | 2

2. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Up to 30 days following the last dose of study drug (Up to 46 days)
Population: The AST population consisted of all Part 1 participants who received at least one dose of study drug (MK-8777 or Placebo).
Measure: Number; unit: participants
Arm/Group | Part 1: Block A MK-8777 | Part 1: Block A Placebo | Part 1: Block B MK-8777 | Part 1: Block B Placebo | Part 1: Block C MK-8777 | Part 1: Block C Placebo | Part 1: Block D MK-8777 | Part 1: Block D Placebo
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With AEs Leading to Discontinuation of Study Drug
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Discontinuation refers to discontinuation of study drug (MK-8777 or Placebo).
Time Frame: Up to the last dose of study drug (Up to 16 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Part 1: Block A MK-8777 | Part 1: Block A Placebo | Part 1: Block B MK-8777 | Part 1: Block B Placebo | Part 1: Block C MK-8777 | Part 1: Block C Placebo | Part 1: Block D MK-8777 | Part 1: Block D Placebo
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 2: Number of Participants With AEs
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product.
Time Frame: Up to 7 days following the last dose of study drug (Up to 35 days)
Population: The AST population consisted of all Part 2 participants who received at least one dose of study drug (MK-8777 or Placebo).
Measure: Number; unit: participants
Arm/Group | Part 2: MK-8777 200 mg | Part 2: MK-8777 800 mg | Part 2: Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants | 10 | 9 | 9

5. Primary Outcome: Part 2: Number of Participants With AEs Leading to Discontinuation of Study Drug
Description: as for outcome 3
Time Frame: Up to the last dose of study drug (Up to 28 days)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Part 2: MK-8777 200 mg | Part 2: MK-8777 800 mg | Part 2: Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants | 0 | 0 | 1

6. Secondary Outcome: Part 1: Change From Baseline in the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item scale designed to assess the severity of depression. The questionnaire includes questions on the following symptoms: Apparent sadness, Reported sadness, Inner tension, Reduced sleep, Reduced appetite, Concentration difficulties, Lassitude, Inability to feel, Pessimistic thoughts, and Suicidal thoughts. Each of the 10 symptoms are rated on a scale of 1 to 6, with 1=absent to 6=severe. The MADRS score can range from 0 (symptoms absent) to 60 (severe depression), with a higher score indicating more severe depression.
Time Frame: Baseline and end of treatment (Up to Day 16)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 1: Block A MK-8777 | Part 1: Block A Placebo | Part 1: Block B MK-8777 | Part 1: Block B Placebo | Part 1: Block C MK-8777 | Part 1: Block C Placebo | Part 1: Block D MK-8777 | Part 1: Block D Placebo
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
score on a scale | -10.00 (7.53) | -24.50 (2.12) | -13.50 (14.46) | -7.00 (8.49) | -10.25 (9.36) | -9.50 (3.54) | -19.00 (9.76) | -2.00 (5.66)

7. Secondary Outcome: Part 2: Change From Baseline in the MADRS
Description: as for outcome 6
Time Frame: Baseline and end of treatment (Up to Day 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: MK-8777 200 mg | Part 2: MK-8777 800 mg | Part 2: Placebo
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | -15.40 (6.40) | -13.70 (11.57) | -13.30 (9.04)

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug for serious AEs (up to 46 days for Part 1; up to 58 days for Part 2). Up to 7 days after last dose of study drug for non-serious AEs (up to 23 days for Part 1; up to 35 days for Part 2).
Arm/Group | Part 1: Block A MK-8777 | Part 1: Block A Placebo | Part 1: Block B MK-8777 | Part 1: Block B Placebo | Part 1: Block C MK-8777 | Part 1: Block C Placebo | Part 1: Block D MK-8777 | Part 1: Block D Placebo | Part 2: MK-8777 200 mg | Part 2: MK-8777 800 mg | Part 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 4/4 | 2/2 | 4/4 | 1/2 | 4/4 | 2/2 | 10/10 | 9/10 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Block A MK-8777 (N=4) | Part 1: Block A Placebo (N=2) | Part 1: Block B MK-8777 (N=4) | Part 1: Block B Placebo (N=2) | Part 1: Block C MK-8777 (N=4) | Part 1: Block C Placebo (N=2) | Part 1: Block D MK-8777 (N=4) | Part 1: Block D Placebo (N=2) | Part 2: MK-8777 200 mg (N=10) | Part 2: MK-8777 800 mg (N=10) | Part 2: Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Colour blindness (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered visual depth perception (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 2 (2) | 1 (1) | 4 (14) | 0 (0) | 2 (2) | 1 (1) | 3 (7) | 3 (4) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling drunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradykinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 2 (2) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (5) | 1 (2) | 2 (3) | 1 (1) | 4 (7) | 0 (0) | 3 (9) | 2 (5) | 5 (8) | 4 (4) | 5 (8)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 3 (4) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 5 (5) | 5 (5)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depersonalisation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phonophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less